CLINICAL TRIAL: NCT01194180
Title: A Phase 1 Study to Evaluate a BCG Challenge Model as a Method of Assessing Anti-mycobacterial Immunity Induced by BCG and a Candidate TB Vaccine, MVA85A, Alone and in Combination
Brief Title: A BCG Challenge Model Study to Assess Anti-mycobacterial Immunity Induced by BCG and a Candidate TB Vaccine, MVA85A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB023
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2011-10

CONDITIONS: Tuberculosis
Keywords: Mycobacterium tuberculosis; BCG; MVA85A
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): BCG-naive subjects receiving intradermal "challenge" injection of BCG and challenge site punch biopsy
  Interventions: Biological: BCG: 100 microlitres ~ 2-8 x 105 pfu
- Group B (Experimental): BCG-naïve subjects receiving intradermal injection of MVA85A followed by intradermal "challenge" injection of BCG and challenge site punch biopsy
  Interventions: Biological: MVA85A: 1 x 108 pfu BCG: 100 microlitres ~ 2-8 x 105 pfu
- Group C (Experimental): BCG-experienced subjects receiving intradermal "challenge" injection of BCG and challenge site punch biopsy
  Interventions: Biological: BCG: 100 microlitres ~ 2-8 x 105 pfu
- Group D (Experimental): BCG-experienced subjects receiving intradermal injection of MVA85A followed by intradermal "challenge" injection of BCG and challenge site punch biopsy
  Interventions: Biological: MVA85A: 1 x 108 pfu BCG: 100 microlitres ~ 2-8 x 105 pfu

INTERVENTIONS:
Biological: BCG: 100 microlitres ~ 2-8 x 105 pfu — BCG vaccination at day C (challenge day) then punch biopsy at day C+14
  Arms: Group A; Group C
Biological: MVA85A: 1 x 108 pfu BCG: 100 microlitres ~ 2-8 x 105 pfu — MVA85A vaccination at day C-28 followed by BCG vaccination at day C (challenge day) then biopsy at day C+14
  Arms: Group B; Group D

SUMMARY:
The purpose of this study is to evaluate the BCG 'challenge' model a four-arm study design has been chosen. Twelve subjects will be recruited into each arm of the study. Allocation of BCG-naïve volunteers to either group A or B, and BCG-vaccinated volunteers to either group C or D, will be performed on a one-to-one alternating basis. Subjects in each group will be challenged by BCG administered intradermally. Prior to challenge, pre-existing immunity to TB will be induced by vaccination with BCG, MVA85A, and both in combination (when compared to BCG- & MVA85A-naïve individuals). BCG quantification will be assessed by analysing the tissue obtained in a punch biopsy of volunteers' skin over the site of BCG 'challenge' vaccination. Any reduction in BCG quantification between groups will then be correlated to existing (and future) laboratory assays of vaccine-induced immune responses in order to identify potential immunological correlates of protection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-55 years
* Resident in or near Oxford for the duration of the study period
* No relevant findings in medical history or on physical examination
* Willingness to allow the Investigators to discuss the individual's medical history with their GP
* Willingness to use effective contraception for the duration of the study period (females only)
* Agreement to refrain from blood donation during the course of the study
* Willingness to give written informed consent
* Agreement to allow the Investigator to register volunteer details with a confidential database to prevent concurrent entry into clinical trials
* Able and willing (in the Investigator's opinion) to comply with all the study requirements

Additional criteria to be met for subjects in group A:

* None

Additional criteria to be met for subjects in group B:

* Willingness to use continuous effective barrier contraception for three months after receiving
* MVA85A vaccination (males and females)

Additional criteria to be met for subjects in group C:

* Confirmation of prior vaccination with BCG not less than three months prior to projected study enrolment date (by visible BCG scar on examination or written documentation)

Additional criteria to be met for subjects in group D:

* Confirmation of prior vaccination with BCG not less than three months prior to projected study enrolment date (by visible BCG scar on examination or written documentation)
* Willingness to use continuous effective barrier contraception for three months after receiving MVA85A vaccination (males and females)

Exclusion Criteria:

* Clinical, radiological, or laboratory evidence of current active TB disease
* Laboratory evidence at screening of latent M. tb infection as indicated by a positive ELISPOT test (>17 sfc/million PBMC) in any ESAT6 peptide or CFP10 peptide poola
* Previous vaccination with candidate TB vaccine MVA85A or candidate TB vaccine FP85A
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* History of serious psychiatric condition
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the study vaccine
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the volunteer in the studyb
* Positive HBsAg, HCV or HIV antibodies
* Female currently lactating, confirmed pregnancy or intention to become pregnant during study period
* Use of an investigational medicinal product or non-registered drug, live vaccine, or medical device other than the study vaccine for 60 days prior to dosing with the study vaccine, or planned use during the study period
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the volunteer at risk or may influence the result of the study or may affect the volunteer's ability to participate in the study

Additional exclusion criteria for subjects in group A:

* Previous vaccination with BCG

Additional exclusion criteria for subjects in group B:

* Previous vaccination with a recombinant MVA vaccine other than MVA85A or FP85A
* Previous vaccination with BCG

Additional exclusion criteria for subjects in group C:

* None

Additional exclusion criteria for subjects in group D:

* Previous vaccination with a recombinant MVA vaccine other than MVA85A or FP85A

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Culture and RT-PCR quantification of BCG in challenge site biopsy | 10 weeks post biopsy

SECONDARY OUTCOMES:
Established and exploratory markers of cell mediated immunity in blood samples and biopsied tissue | 10 weeks post biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxon, United Kingdom

REFERENCES:
- [Derived] Tanner R, Satti I, Harris SA, O'Shea MK, Cizmeci D, O'Connor D, Chomka A, Matsumiya M, Wittenberg R, Minassian AM, Meyer J, Fletcher HA, McShane H. Tools for Assessing the Protective Efficacy of TB Vaccines in Humans: in vitro Mycobacterial Growth Inhibition Predicts Outcome of in vivo Mycobacterial Infection. Front Immunol. 2020 Jan 10;10:2983. doi: 10.3389/fimmu.2019.02983. eCollection 2019. PMID 31998295
- [Derived] Harris SA, Meyer J, Satti I, Marsay L, Poulton ID, Tanner R, Minassian AM, Fletcher HA, McShane H. Evaluation of a human BCG challenge model to assess antimycobacterial immunity induced by BCG and a candidate tuberculosis vaccine, MVA85A, alone and in combination. J Infect Dis. 2014 Apr 15;209(8):1259-68. doi: 10.1093/infdis/jit647. Epub 2013 Nov 23. PMID 24273174